CLINICAL TRIAL: NCT03082547
Title: A Clinical Observation on Neuropsychology and Electrophysiology in Headache Patinets With Myofascial Trigger Points
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qi Wan, chief physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: myofascial trigger points
Record Dates: First submitted 2017-03-04; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Myofascial Trigger Points
Keywords: Headache; Neuropsychological tests; Myofascial trigger points; electrophysiology
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Headache Groub: Headache patients with myofascial trigger points.
- Healthy Groub: No headache or other diseases can cause headaches of healthy people.

SUMMARY:
To study the clinical characteristics of headache patients with pericranial myofascial trigger points(MTrPs),and to explore the possible pathogenesis of MTrPs,investigators hope to find the possible electrical biomarkers for clinical diagnosis and treatment, and to improve the effect of headache treatment.

DETAILED DESCRIPTION:
A series of neuropsychological test scale including Mini-mental State Examination(MMSE),Hamilton Anxiety Rating Scale(HAMA) and Hamilton Depression Rating Scale (HMAD) were evaluated among all patients.The needle pole electromyography (EMG) inspection were practiced on subjects with myofascial trigger points ,for analysing those electrophysiological characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Primary headache patients with pericranial myofascial trigger points.

Exclusion Criteria:

* Cranial weeks muscle infection or trauma, medical history, physical examination, laboratory and imaging studies suggest secondary headache patients except cervicalheadache.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: To enroll headache patients with pericranial myofascial trigger points into the groups in our hospital outpatients and inpatients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Electromyography | 30 minutes
  The needle pole electromyography (EMG) inspection

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale(HAMA) | 20 minutes
  Evaluating Anxiety state: Total score without anxiety symptoms less than 7 ,> 7 points might be anxious, > 14 points must be anxious, > 21 points obvious anxiety, 29 > serious anxiety
Mini-mental State Examination(MMSE) | 20 minutes
  Evaluating cognitive State, MMSE boundary between normal and abnormal value related to the degree of education, literacy (not education) group of 17 points or less, primary school (education duration of 6 years or less) group of 20 or less, secondary or above (education duration of > 6 years) group of 24 points or less, the following boundary value for cognitive function defect, above normal.
Hamilton Depression Rating Scale (HMAD) | 20 minutes
  Evaluating depression state:Normal score < 8 points, 8 ~ 20 points might be depression, 20 ~ 35 must have depression, > 35 severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The needle pole electromyography, Nanjing, Jiangsu, China